CLINICAL TRIAL: NCT00399165
Title: Oral Androgens in Man-4: Gonadotropin Suppression Medicated by Oral Testosterone Enanthate in Oil Plus Dutasteride (Short Title: Oral T-4)
Brief Title: Oral Androgens in Man-4: (Short Title: Oral T-4)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: John K Amory, MD, MPH, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 06-2962-A; U54HD042454 (NIH); K23HD045386 (NIH)
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Contraception
Keywords: Oral Contraception for Men; Contraceptive agent
MeSH Terms: interventions — testosterone enanthate; Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Oral Testosterone enanthate in sesame oil, 400 mg po (orally), BID (twice daily) + dutasteride 0.5 mg orally, qd (once daily) for 28 days + dutasteride load 24.5 mg po once
  Interventions: Drug: Testosterone Enanthate; Drug: Dutasteride
- 2 (Active Comparator): Oral Testosterone sesame oil, 800 mg po (orally), qd (in am daily) + placebo sesame oil (in pm daily) + dutasteride 0.5 mg orally, qd (once daily) for 28 days + dutasteride load 24.5 mg po once
  Interventions: Drug: Testosterone Enanthate; Drug: Dutasteride; Other: placebo sesame oil

INTERVENTIONS:
Drug: Testosterone Enanthate — Oral Testosterone 400 mg orally for 28 days
  Other Names: Delatestryl
  Arms: 1
Drug: Testosterone Enanthate — Oral Testosterone 800 mg orally for 28 days
  Other Names: Delatestryl
  Arms: 2
Drug: Dutasteride — dutasteride 0.5 mg orally, once daily for 28 days
  Other Names: Avodart
Other: placebo sesame oil — placebo sesame oil
  Arms: 2
Drug: Dutasteride — 24.5 mg po once (Day 0)
  Other Names: Avodart

SUMMARY:
The protocol was designed to address the hypothesis that oral testosterone enanthate plus dutasteride can suppress the secretion of LH and FSH after four weeks of administration. In addition, we will compare the gonadotropin suppression mediated by a dose of testosterone enanthate (400 mg twice daily) that would be expected to maintain the serum testosterone in the normal range throughout the day, with the same dose (800 mg once daily) administered once daily. This larger once-daily dose is expected to result in a higher peak and lower trough by the end of the dosing interval

DETAILED DESCRIPTION:
This study will be carried out in a double-blinded fashion, so neither the subject nor the investigator will be aware of treatment assignment during the study. This protocol is designed to address the hypothesis that oral testosterone enanthate plus dutasteride can suppress the secretion of LH and FSH after four weeks of administration. In addition, we will compare the gonadotropin suppression mediated by a dose of testosterone enanthate (400 mg twice daily) that would be expected to maintain the serum testosterone in the normal range throughout the day, with the same dose (800 mg once daily) administered once daily. This larger once-daily dose is expected to result in a higher peak and lower trough by the end of the dosing interval. Secondary endpoints in this study include the ability of oral testosterone enanthate plus dutasteride to maintain short-term androgen-mediated endpoints such as mood and sexual function over the 4-week treatment period as well as weekly measures of safety, including blood counts, PSA and liver and kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 to 55 years of age
* In good general health based on normal screening evaluation (consisting of a medical history, physical exam, normal serum chemistry, hematology, and baseline hormone levels)
* Subject must agree not to participate in another research drug study for the duration of the study
* Subject must agree to not donate blood during the study
* Subject must be willing to comply with the study protocol and procedures

Exclusion Criteria:

* Men in poor general health, with abnormal blood results (clinical laboratory tests or hormone values)
* A known history of alcohol or drug abuse
* A history of testicular disease or severe testicular trauma,
* A history of bleeding disorders or current use of anti-coagulants
* A history of sleep apnea and/or major psychiatric disorders
* A body-mass index greater than 35,
* A history of or current use of testosterone
* Infertility

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Dutasteride can suppress the secretion of LH and FSH after four weeks of administration. | 4 weeks

SECONDARY OUTCOMES:
The ability of oral testosterone enanthate plus dutasteride to maintain short-term androgen-medicated endpoints such as mood and sexual function over the 4-week treatment period | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Martin CW, Anderson RA, Cheng L, Ho PC, van der Spuy Z, Smith KB, Glasier AF, Everington D, Baird DT. Potential impact of hormonal male contraception: cross-cultural implications for development of novel preparations. Hum Reprod. 2000 Mar;15(3):637-45. doi: 10.1093/humrep/15.3.637. PMID 10686211
- [Background] Weston GC, Schlipalius ML, Bhuinneain MN, Vollenhoven BJ. Will Australian men use male hormonal contraception? A survey of a postpartum population. Med J Aust. 2002 Mar 4;176(5):208-10. doi: 10.5694/j.1326-5377.2002.tb04374.x. PMID 11999235
- [Background] Heinemann K, Saad F, Wiesemes M, White S, Heinemann L. Attitudes toward male fertility control: results of a multinational survey on four continents. Hum Reprod. 2005 Feb;20(2):549-56. doi: 10.1093/humrep/deh574. Epub 2004 Dec 17. PMID 15608042
- [Background] Amory JK, Bremner WJ. Oral testosterone in oil plus dutasteride in men: a pharmacokinetic study. J Clin Endocrinol Metab. 2005 May;90(5):2610-7. doi: 10.1210/jc.2004-1221. Epub 2005 Feb 15. PMID 15713724
- [Background] Amory JK, Page ST, Bremner WJ. Oral testosterone in oil: pharmacokinetic effects of 5alpha reduction by finasteride or dutasteride and food intake in men. J Androl. 2006 Jan-Feb;27(1):72-8. doi: 10.2164/jandrol.05058. PMID 16400081
- [Background] Bebb RA, Anawalt BD, Christensen RB, Paulsen CA, Bremner WJ, Matsumoto AM. Combined administration of levonorgestrel and testosterone induces more rapid and effective suppression of spermatogenesis than testosterone alone: a promising male contraceptive approach. J Clin Endocrinol Metab. 1996 Feb;81(2):757-62. doi: 10.1210/jcem.81.2.8636300.
- [Background] Anawalt BD, Bebb RA, Bremner WJ, Matsumoto AM. A lower dosage levonorgestrel and testosterone combination effectively suppresses spermatogenesis and circulating gonadotropin levels with fewer metabolic effects than higher dosage combinations. J Androl. 1999 May-Jun;20(3):407-14. PMID 10386821
- [Background] Anawalt BD, Amory JK, Herbst KL, Coviello AD, Page ST, Bremner WJ, Matsumoto AM. Intramuscular testosterone enanthate plus very low dosage oral levonorgestrel suppresses spermatogenesis without causing weight gain in normal young men: a randomized clinical trial. J Androl. 2005 May-Jun;26(3):405-13. doi: 10.2164/jandrol.04135. PMID 15867009
- [Result] Amory JK, Kalhorn TF, Page ST. Pharmacokinetics and pharmacodynamics of oral testosterone enanthate plus dutasteride for 4 weeks in normal men: implications for male hormonal contraception. J Androl. 2008 May-Jun;29(3):260-71. doi: 10.2164/jandrol.107.004226. Epub 2007 Nov 28. PMID 18046048